CLINICAL TRIAL: NCT04472143
Title: Granisetron Transdermal Delivery System for Prophylaxis of Nausea and Vomiting in Patients Receiving Oral Anticancer Agents: a Single-center, Single-arm, Phase II Trial
Brief Title: Granisetron Transdermal Patch for Prophylaxis of Nausea and Vomiting in Patients Receiving Oral Anticancer Agents
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SS-SP01-201904
Record Dates: First submitted 2020-07-02; First posted 2020-07-15 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Chemotherapy-induced Nausea and Vomiting (CINV)
Keywords: oral anticancer agents
MeSH Terms: conditions — Vomiting | interventions — Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Granisetron Transdermal Delivery System (Experimental): The patch will be applied to the upper arm 24-48 hours before the start of chemotherapy, and left in place for 7 days
  Interventions: Drug: Granisetron Transdermal Delivery System

INTERVENTIONS:
Drug: Granisetron Transdermal Delivery System — A total of 60 patients with HER2-positive advanced breast cancer who are scheduled to receive pirotinib combined with capecitabine will be enrolled. A single transdermal patch will be applied to the subject' upper outer arm 24-48 hours before chemotherapy for 7 days. The observation period will be from the time of enrollment to 14 days (± 7 days) after the removal of granisetron patch.
  Other Names: sancuso; granisetron transdermal patch

SUMMARY:
At present, the clinical studies of 5-HT3RA are aimed at nausea and vomiting induced by single-day chemotherapy, but there are many chemotherapy schemes that require multi-day administration in clinical practice. Compared with single-day chemotherapy, multi-day chemotherapy (including multi-day intravenous chemotherapy and multi-day administration of oral antineoplastic drugs) faces a more complex situation, requiring the prevention of both acute CINV, and delayed CINV at the same time. Clinically, oral or intravenous 5-HT3 antagonists are needed for many times, and the convenience is poor. Especially with the increasing application of oral antineoplastic drugs (including oral chemotherapeutic drugs and oral molecular targeted drugs), the nausea and vomiting caused by oral antineoplastic drugs have attracted more and more attention of clinicians. Pyrotinib is an oral, irreversible pan-ErbB receptor tyrosine kinase inhibitor (TKI) with activity against epidermal growth factor receptor (EGFR)/HER1, HER2, and HER4.12 Preclinical data suggest that pyrotinib can irreversibly inhibit multiple ErbB receptors and effectively inhibit the proliferation of HER2-overexpressing cells both in vivo and in vitro. Pirotinib is an effective drug that progresses after treatment with trastuzumab. At present, pirrotinib combined with capecitabine has made a major breakthrough in the treatment of recurrent and metastatic HER-positive breast cancer, with a median PFS of 18.1 months and an ORR of 78.5%. Although most adverse reactions are controllable, the program The incidence of related nausea and vomiting has reached about 50%, and nausea and vomiting most often occurred in the first week after treatment, which not only affected the patient's quality of life, but also affected the treatment compliance of the two oral drugs to a certain extent. It has become a more difficult problem for clinicians in the treatment process.

DETAILED DESCRIPTION:
Chemotherapy-induced nausea and vomiting (CINV) are commonly occurring, which have a negative impact on patient's quality of life and lead to poor compliance with further chemotherapy. In addition, nausea and vomiting can result in dehydration, electrolyte imbalances, anorexia and malnutrition, further withdrawal from treatment. Thus, the prevention of CINV could be one of the most challenging supportive care issues in oncology.

The development of the 5-HT3-receptor antagonists (5-HT3RA, i.e., granisetron, ondansetron) represents a significant advance in antiemetic therapy. All of these agents show considerable efficacy in preventing CINV, with acute responses for single agents ranging from 40% to 86%. The granisetron transdermal delivery system (GTDS;Sancuso®, ProStrakan, Inc., USA) has been recently developed and approved by the US Food and Drug Administration (FDA) for prevention and controlling of CINV. Sancuso® is the first GTDS for prevention and control of CINV, which contain 34.3 mg of granisetron and can provide continuous delivery of granisetron through the skin, with releasing 3.3 mg of granisetron per 24 h for up to 7 days. Meanwhile, it maintained the plasma concentration (Cavg) of 2.2 ng/mL over 6 days, similar to that obtained with 2 mg of oral granisetron administered every day during the same period of time. Compared with other 5-HT3RAS, GTDS carries important advantages over repeated injections or oral dosing in terms of patient convenience and compliance. It may be especially valuable in patients for whom swallowing is difficult or absorption of oral medication is uncertain, such as cancer patients with gastrointestinal surgery.

At present, the clinical studies of 5-HT3RA are aimed at nausea and vomiting induced by single-day chemotherapy, but there are many chemotherapy schemes that require multi-day administration in clinical practice. Compared with single-day chemotherapy, multi-day chemotherapy (including multi-day intravenous chemotherapy and multi-day administration of oral antineoplastic drugs) faces a more complex situation, requiring the prevention of both acute CINV, and delayed CINV at the same time. Clinically, oral or intravenous 5-HT3 antagonists are needed for many times, and the convenience is poor. Especially with the increasing application of oral antineoplastic drugs (including oral chemotherapeutic drugs and oral molecular targeted drugs), the nausea and vomiting caused by oral antineoplastic drugs have attracted more and more attention of clinicians. Pyrotinib is an oral, irreversible pan-ErbB receptor tyrosine kinase inhibitor (TKI) with activity against epidermal growth factor receptor (EGFR)/HER1, HER2, and HER4.12 Preclinical data suggest that pyrotinib can irreversibly inhibit multiple ErbB receptors and effectively inhibit the proliferation of HER2-overexpressing cells both in vivo and in vitro. Pirotinib is an effective drug that progresses after treatment with trastuzumab. At present, pirrotinib combined with capecitabine has made a major breakthrough in the treatment of recurrent and metastatic HER-positive breast cancer, with a median PFS of 18.1 months and an ORR of 78.5%. Although most adverse reactions are controllable, the program The incidence of related nausea and vomiting has reached about 50%, and nausea and vomiting most often occurred in the first week after treatment, which not only affected the patient's quality of life, but also affected the treatment compliance of the two oral drugs to a certain extent. It has become a more difficult problem for clinicians in the treatment process.

A published phase III trial (392MD/15/C) in 641 patients receiving multiday moderately emetogenic chemotherapy (MEC) or highly emetogenic chemotherapy (HEC) regimen demonstrated that the GTDS was not inferior to oral granisetron in complete control (CC) of CINV. Though 71% of patients included in the GTDS group received cisplatin-based HEC and without the use of neurokinin-1 (NK-1) RA, the efficacy was satisfying and promising. Only 11.9% of Asian patients were included in the study and 43 Asian patients was administrated GTDS.

A randomized, active control, double-blind, parallel-group study, conducted at 15 centers in China. The primary objective was to demonstrate GTDS efficacy compared to oral granisetron in Chinese patients. Secondary objectives included the assessment of the safety, tolerability and adhesive properties of the GTDS. Patients were randomized in a 1:1 ratio using a central randomization system to receive either a GTDS patch and placebo tablets or a placebo patch and active tablets (1 mg granisetron). Stratification was based on gender, the severity of emetogenic chemotherapy (moderate or high risk) and chemotherapy duration (2 or ≥3d). The primary efficacy endpoint was the percentage of patients achieving complete control of CINV (CC; no vomiting and/or retching, no more than mild nausea, and no need for rescue medication) from the first administration until 24 h after the last administration of chemotherapeutic agents (PEEP). The CC of per day (day 1, 2, 3, 4, 5) during PEEP was observed. Secondary efficacy endpoints were the following: the time to failure of CC during the efficacy observation period (the chemotherapy initiation until 24 h after patch removal), the percentage of patients failing CC due to nausea, vomiting, or receipt of rescue medication (total days and per day), the percentage of patients achieving complete response (CR; no vomiting and/or retching, no use of rescue medication) during PEEP, patients' global satisfaction with antiemetic therapy (assessed using a 10-cm visual analog scale (VAS) at the time of patch removal), the frequency of vomiting per day and the severity of nausea during the efficacy observation period, and the percentage adhesion of the patch over the application period. Further analyses showed that the difference of CC percentage occurred on the first day of chemotherapy between the groups. In the FAS, the CC percentage of CINV was 70.13% in the GTDS group and 91.03% in the oral granisetron group on day 1 of chemotherapy. Statistical significance was observed (P<0.0001). But in the following day 2 to day 5, the CC remained stable lever in the GTDS group (69.48-79.63%). While in the oral granisetron group, the CC decreased to 76.3% on day 2 and then remained the similar level from day 3 to day 5 (67.26-76.28%). Overall, the percentage CC of CINV was similar and there was no statistical significance in both groups (P>0.05). The same conclusion was also drawn from the PPS analyses. The predefined subgroups analyses included chemotherapy duration, sex, cisplatin-contained in the chemotherapy regimen and smoking history.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged ≥ 18 years;
2. Histologically and/or cytologically confirmed locally advanced/metastatic breast cancer;
3. The physical status score ECOG ≤ 2；
4. Life expectancy of ≥3 months;
5. Will receive the first treatment cycle of oral pirotinib combined with capecitabine;
6. In accordance with the indication of chemotherapy and basic requirements;

   * Peripheral haematology: Hb ≥9.0g/dL; absolute neutrophil count ≥1.5×109/L；platelet count ≥80×109/L
   * Blood biochemistry: Total bilirubin < 1.25×ULN, ALT and AST ≤ 2.5×ULN; if liver metastasis, ALT and AST < 5×ULN, Creatinine ≤ 1×ULN, basic normal serum electrolyte (Na, Ka, Cl, Ca)
   * Other important organs function normally
7. Subjects voluntarily participate and signed the informed consent form.

Exclusion Criteria:

1. Contraindicated to 5-HT receptor antagonists (such as gastrointestinal obstruction) or allergy to 5-HT;
2. Any nausea and vomiting (II or above) within 72 hours before the start of chemotherapy;
3. Liver and kidney diseases, infections, and diseases of central nervous system or mental health. Patients who are evaluated by investigators as unsuitable for inclusion;
4. Prolonged QT interval at baseline (QTc>470msec at baseline);
5. Patients scheduled to receive radiotherapy of whole body, brain or upper abdomen;
6. Confirmed by craniocerebral CT or MRI, patients with brain tumor lesions or patients taking drugs to treat brain tumors or epileptic symptoms;
7. Patens unable to cooperate and describe treatment response;
8. History of drug abuse and alcohol dependence;
9. Pregnancy, lactation or intended pregnancy;
10. History of allergic reactions to drugs with similar chemical structures, or to transdermal therapeutic systems, including commercial dressings such as Elastoplast®
11. Those who have participated or plan to participate in other clinical trials of granisetron; those who have participated in other clinical trials within 30 days before enrollment;
12. Unable to eat for any reason;
13. Other situations evaluated by investigators as unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-07-18 (Actual); Primary Completion 2022-09-18 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects achieving complete response of nausea and vomiting (complete response is defined as no vomiting and/or retching, and no rescue medication) within 7 days after administration | 7 days
  complete response means no vomiting, and no rescure medication (day 1-7)

SECONDARY OUTCOMES:
The percentage of subjects achieving complete response of nausea and vomiting on days 1-3 (acute phase) and on days 4-7 (delayed phase) after administration | 7 days
  complete response means no vomiting, and no rescure medication
The percentage of subjects achieving complete control of nausea and vomiting (complete control is defined as no vomiting and/or retching, no more than mild nausea, and no rescue medication) within 7 days after administration | 7 days
  complete control means no vomiting, mild nausea and no rescue medication
The percentage of subjects achieving complete control of nausea and vomiting on days 1-3 (acute phase) and on days 4-7 (delayed phase) after administration | 7 days
  complete control means no vomiting, mild nausea and no rescure medication (day 1-3)
Patients' satisfaction with antiemetic therapy (assessed using a 10-cm visual analog scale at the time of patch removal） | 7 days
  "dissatisfied" on the left end (0 cm) of visual analog scale and the "very satisfied"on the right end of visual analog scale (10 cm)
The frequency of vomiting episodes per day after the administration of oral chemotherapy during the observation period (the oral chemotherapy initiation until 24 h after patch removal) | 7 days
  the number of vomiting each day will be recored by patients
Severity of nausea per day during the observation period (the oral chemotherapy initiation until 24 h after patch removal) | 7 days
  the degree of nausea each day will be recored by patients

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, Prof., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coluzzi F, Mattia C. Management of chemotherapy-induced nausea and vomiting in patients receiving multiple-day highly or moderately emetogenic chemotherapy: role of transdermal granisetron. Future Oncol. 2016 Aug;12(16):1865-76. doi: 10.2217/fon-2016-0097. Epub 2016 May 17. PMID 27184113
- [Background] Navari RM, Aapro M. Antiemetic Prophylaxis for Chemotherapy-Induced Nausea and Vomiting. N Engl J Med. 2016 Apr 7;374(14):1356-67. doi: 10.1056/NEJMra1515442. No abstract available. PMID 27050207